CLINICAL TRIAL: NCT02294162
Title: Pain Relief for Submucosal Resection of Nasal Septum in Adults Does Ketamine Have a Pre-Emptive Effect?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by IRB
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Ronen Ohad, MD,, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0104-14
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5 mg/kg body weight Ketamin (Experimental): Patients allocated to this arm will receive an iv dose of 0.5 mg/kg body weight ketamine.
  Interventions: Drug: Ketamine i.v
- 5 ml normal saline as placebo (Placebo Comparator): Patients allocated to this arm will receive an iv dose of 5ml saline as placebo.
  Interventions: Drug: Ketamine i.v

INTERVENTIONS:
Drug: Ketamine i.v

SUMMARY:
Pain is an unpleasant sensory experience associated with actual or potential tissue damage. Acute pain management is an important aspect of perioperative anesthetic care. Moreover, it is the most important factor related to patient discomfort after surgery. Adequate pain management, ideally resulting in the complete absence of postoperative pain, not only provides comfort to patients, but may also contribute to improved healing and a reduction in the incidence of postoperative complications. Inadequate postoperative analgesia has been shown to contribute to adverse outcomes, including, but not limited to, immunosuppression, hyperglycemia, poor rehabilitation, and progression to chronic pain.

DETAILED DESCRIPTION:
Patients who are scheduled for submucosal resection of nasal septum with or without turbinectomy will be recruited for the study The patients will be will be assigned to either the treatment group who will be administered ketamine prior to the operation or the control group who will receive a normal saline injection, both in identicle syringes.

All patients will be operated on by the same surgoens and by the same method of dissection and hemostasis (2-5 2 ml lidocadrain carpules, monopolar suction-cautery set on 25).

Patients folow-up will be reported in their medical charts. The post operative analgetic effect will be assessed by the amount of analgesia required in the post-operative period and by regular pain measurements using VAS (Visual Analogue Scale) - at 0.5 hours post operation in the recovery room, 8 hours post operation and the morning of first post operative day in the otolaryngology - head and neck department

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing submucosal resection of nasal septum with or without turbinectomy.
* Over 18 years of age.
* ASA (anesthsiology Severity Score) score of 1-2.
* Signed informed consent by patient or caregiver.

Exclusion Criteria:

* Allergy to Ketamine
* Unable/ unwilling to comply with the protocol requirements
* Pregnancy or breast feeding
* Chronic use of analgetics
* History of alcohol and/or drug abuse
* Previous nasal surgry

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Pain: reduction in severity based on VAS score. | the morning of first post operative day
  The post operative analgetic effect will be assessed by the amount of analgesia required in the post-operative period and by regular pain measurements using VAS (Visual Analogue Scale) - at 0.5 hours post operation in the recovery room, 8 hours post operation and the morning of first post operative day
consumption of postoperative pain medication type, dosage and reduction in the demand postoperatively. | the morning of first post operative day
  The data will be collected from the medical file

SECONDARY OUTCOMES:
Readmission for any reason. | one week
Duration of hospital stay. | one week

CONTACTS AND LOCATIONS:
Locations (1):
- Galillee medical center, Nahariya, Israel